CLINICAL TRIAL: NCT01623167
Title: Eltrombopag Added to Standard Immunosuppression in Treatment-Naive Severe Aplastic Anemia
Brief Title: Eltrombopag With Standard Immunosuppression for Severe Aplastic Anemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120150; 12-H-0150
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Severe Aplastic Anemia
Keywords: Pancytopenia; Immunosuppression; Hematopoesis; Autoimmunity; Thrombocytopenia
MeSH Terms: conditions — Anemia, Aplastic; Pancytopenia; Autoimmune Diseases; Thrombocytopenia | interventions — Cyclosporine; eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: hATG, CsA, EPAG Day 14 to Month 6 (Experimental): Receive horse ATG days 1- 4, receive CsA day 1 to month 6, and receive eltrombopag day 14 to month 6
  Interventions: Drug: Cohort 1: hATG, CsA, EPAG Day 14 to Month 6
- Cohort 2: hATG, CsA, EPAG Day 14 to Month 3 (Experimental): Receive horse ATG days 1- 4, receive CsA day 1 to month 6, and receive eltrombopag day 14 to month 3
  Interventions: Drug: Cohort 2: hATG, CsA, EPAG Day 14 to Month 3
- Cohort 3: hATG, CsA (dose reduced), EPAG day 1 to month 6 (Experimental): Receive horse ATG days 1- 4, receive CsA day 1 to month 6 at higher dose, then reduced dose for 18months, and receive eltrombopag day 1 to month 6
  Interventions: Drug: Cohort 3: hATG, CsA (dose reduced), EPAG day 1 to month 6
- Extrension Cohort (Experimental): Receive horse ATG days 1- 4, receive CsA day 1 to month 6 at higher dose, then reduced dose for 18 months, and receive eltrombopag day 1 to month 6
  Interventions: Drug: Extension Cohort

INTERVENTIONS:
Drug: Cohort 1: hATG, CsA, EPAG Day 14 to Month 6 — hATG (standard of care) administered for 4 days, CsA (standard of care) administered starting day 1 for 6 months, eltrombopag (experimental) administered Day 14 to month 6
  Other Names: Horse Antithymocyte Globulin, Cyclosporine, Promacta, Eltrombopag
  Arms: Cohort 1: hATG, CsA, EPAG Day 14 to Month 6
Drug: Cohort 2: hATG, CsA, EPAG Day 14 to Month 3 — hATG (standard of care) administered for 4 days, CsA (standard of care) administered starting day 1 for 6 months, eltrombopag (experimental) administered Day 14 to month 3
  Other Names: Horse Antithymocyte Globulin, Cyclosporine, Promacta, Eltrombopag
  Arms: Cohort 2: hATG, CsA, EPAG Day 14 to Month 3
Drug: Cohort 3: hATG, CsA (dose reduced), EPAG day 1 to month 6 — hATG (standard of care) administered for 4 days, CsA (standard of care) administered starting day 1 for 6 months at higher dose, then reduced dose for 18 months, eltrombopag (experimental) administered Day 1 to month 6
  Other Names: Horse Antithymocyte Globulin, Cyclosporine, Promacta, Eltrombopag
  Arms: Cohort 3: hATG, CsA (dose reduced), EPAG day 1 to month 6
Drug: Extension Cohort — Receive horse ATG days 1- 4, receive CsA day 1 to month 6 at higher dose, then reduced dose for 18 months, and receive eltrombopag day 1 to month 6
  Other Names: Horse Antithymocyte Globulin (hATG), Cyclosporine (CsA), Promacta, Eltrombopag (EPAG)
  Arms: Extrension Cohort

SUMMARY:
Background:

* Severe aplastic anemia is a rare and serious blood disorder. It happens when the immune system starts to attack the bone marrow cells. This causes the bone marrow to stop making red blood cells, platelets, and white blood cells. Standard treatment for this disease is horse-ATG and cyclosporine, which suppress the immune system and stop it from attacking the bone marrow. However, this treatment does not work in all people. Some people still have poor blood cell counts even after treatment.
* Eltrombopag is a drug designed to mimic a protein in the body called thrombopoietin. It helps the body to make more platelets. It may also cause the body to make more red and white blood cells. Studies have shown that eltrombopag may be useful when added to standard treatment for severe aplastic anemia. It may help improve poor blood cell counts.

Objectives:

- To test the safety and effectiveness of adding eltrombopag to standard immunosuppressive therapy for severe aplastic anemia.

Eligibility:

- Individuals at least 2 years of age who have severe aplastic anemia that has not yet been treated.

Design:

* Participants will be screened with a physical exam, medical history, and blood tests. Blood and urine samples will be collected.
* Participants will start treatment with horse-ATG and cyclosporine. Treatment will be given according to the standard of care for the disease.
* Cohort 1: After 14 days, participants will start taking eltrombopag. They will take eltrombopag for up to 6 months.
* Cohort 2: After 14 days, participants will start taking eltrombopag. They will take eltrombopag for up to 3 months.
* Cohort 3 and Extension Cohort: Participants will start taking eltrombopag on Day 1. They will take eltrombopag for up to 6 months.
* Participants may receive other medications to prevent infections during treatment.
* Treatment will be monitored with frequent blood tests. Participants will also fill out questionnaires about their symptoms and their quality of life.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and a hypocellular bone marrow. Allogeneic bone marrow transplantation offers the opportunity for cure in younger patients, but most are not suitable candidates for transplantation due to advanced age or lack of a histocompatible donor. Comparable long-term survival in SAA is attainable with immunosuppressive treatment with horse anti-thymocyte globulin (h-ATG) and cyclosporine (CsA). However, of those patients treated with h-ATG/CsA, one quarter to one third will not respond, and 30-40% of responders relapse. The majority of the hematologic responses observed following initial h-ATG/CsA are partial, with only a few patients achieving normal blood counts. Furthermore, analysis of our own extensive clinical data suggests that poor blood count responses to a single course of ATG (non-robust responders), even when transfusion-independence is achieved, predicts a worse prognosis than when robust hematologic improvement is achieved (protocol 90-H-0146). The explanation for partial recovery and relapse are not fully understood, but incomplete elimination of auto-reactive T cells and insufficient stem cell reserve are both possible. Furthermore, 10-15% of SAA patients treated with standard immunosuppression will develop an abnormal karyotype in follow-up, with monosomy 7 being most common, which portends progression to myelodysplasia and leukemia. In contrast, malignant clonal evolution is rare in complete responders to immunosuppression. Although horse ATG/CsA represented a major advance in the treatment of SAA, refractoriness, incomplete responses, relapse, and clonal evolution limit the success of this modality. Thus, newer regimens are needed to address these limitations, and provide a better alternative to stem cell transplantation.

One approach to augment the quality of hematologic responses is to improve underlying stem cell function. Previous attempts to improve responses in SAA with hematopoietic cytokines including erythropoietin, G-CSF, and stem cell factor, have failed. Thrombopoietin (TPO) is the principal endogenous regulator of platelet production. In addition, TPO also has stimulatory effects on more primitive multilineage progenitors and stem cells in vitro and in animal models. Eltrombopag (Promacta ), an oral 2nd generation small molecule TPO-agonist, is currently approved for treatment of chronic immune thrombocytopenic purpura (ITP), chronic hepatitis C-associated thrombocytopenia, and severe aplastic anemia who have had an insufficient response to immunosuppressive therapy. Eltrombopag increases platelets in healthy subjects and in thrombocytopenic patients with chronic ITP and hepatitis C virus (HCV) infection. Our Branch recently completed a pilot study of eltrombopag in refractory SAA. We saw encouraging clinical results in a cohort of patients who have failed on average two prior immunosuppressive regimens (Olnes et al. ASH Annual Meeting Abstracts, San Diego, CA, 2011, oral presentation and N Engl J Med 2012;367:11-9.1). Of the twenty-five SAA patients treated with eltrombopag by mouth for three months, eleven (44%) patients met protocol criteria of clinically meaningful hematologic responses, without significant toxicity. Nine patients demonstrated an improvement in thrombocytopenia (>20k/ L increase or transfusion independence), hemoglobin improved in two patients (>1.5g/dL or achieved transfusion independence, and four patients had a significant response in their neutrophil count. When responders continued the drug beyond three months, the hematologic response to eltrombopag increased; a trilineage response was observed in four patients, and a bilineage response occurred in another four, with median follow-up of 13 months. These results suggest that stem cell depletion, a major component of the pathophysiology of SAA, might be directly addressed by eltrombopag administration. The aim of the current study would be to improve the hematologic response rate and its quality, as well as prevent late complications such as relapse and clonal progression, by addition of eltrombopag to standard immunosuppressive therapy.

This trial will evaluate the safety and efficacy of combining eltrombopag with standard hATG/CSA as first line therapy in patients with SAA. The primary endpoint will be the rate of complete hematologic response at six months. Secondary endpoints are relapse, robust hematologic blood count recovery at 3, 6, and 12 months, survival, clonal evolution to myelodysplasia and leukemia, marrow stem cell content and hematological response of relapse patients that re-start treatment.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Severe aplastic anemia characterized by Bone marrow cellularity less than 30 percent (excluding lymphocytes)

   AND

   At least two of the following:
   * Absolute neutrophil count less than 500/microL
   * Platelet count less than 20,000/microL

   Absolute reticulocyte count less than 60,000/microL
2. Age greater than or equal to 2 years old
3. Weight greater than 12 kg

EXCLUSION CRITERIA:

1. Known diagnosis of Fanconi anemia
2. Evidence of a clonal disorder on cytogenetics performed within 12 weeks of study entry. Patients with super severe neutropenia (ANC less than 200 /microL) will not be excluded initially if cytogenetics are not available or pending. If evidence of a clonal disorder consistent with myelodysplasia is later identified, the patient will go off study.
3. Prior immunosuppressive therapy with any ATG, alemtuzumab, or high dose cyclophosphamide
4. SGOT or SGPT >5 times the upper limit of normal
5. Subjects with known liver cirrhosis in severity that would preclude tolerability of cyclosporine and eltrombopag as evidenced by albumin < 35g/L
6. Hypersensitivity to eltrombopag or its components
7. Infection not adequately responding to appropriate therapy
8. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 7-10 days is likely
9. Potential subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible
10. Current pregnancy, or unwillingness to take oral contraceptives or use a barrier method of birth control or practice abstinence to refrain from pregnancy if of childbearing potential during the course of this study
11. Inability to understand the investigational nature of the study or to give informed consent or does not have a legally authorized representative or surrogate that can provide informed consent.

Ages: 2 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2029-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Zoumbos NC, Gascon P, Djeu JY, Trost SR, Young NS. Circulating activated suppressor T lymphocytes in aplastic anemia. N Engl J Med. 1985 Jan 31;312(5):257-65. doi: 10.1056/NEJM198501313120501. PMID 2981406
- [Background] Young NS, Leonard E, Platanias L. Lymphocytes and lymphokines in aplastic anemia: pathogenic role and implications for pathogenesis. Blood Cells. 1987;13(1-2):87-100. PMID 3311225
- [Background] Townsley DM, Scheinberg P, Winkler T, Desmond R, Dumitriu B, Rios O, Weinstein B, Valdez J, Lotter J, Feng X, Desierto M, Leuva H, Bevans M, Wu C, Larochelle A, Calvo KR, Dunbar CE, Young NS. Eltrombopag Added to Standard Immunosuppression for Aplastic Anemia. N Engl J Med. 2017 Apr 20;376(16):1540-1550. doi: 10.1056/NEJMoa1613878. PMID 28423296
- [Derived] Zaimoku Y, Patel BA, Adams SD, Shalhoub R, Groarke EM, Lee AAC, Kajigaya S, Feng X, Rios OJ, Eager H, Alemu L, Quinones Raffo D, Wu CO, Flegel WA, Young NS. HLA associations, somatic loss of HLA expression, and clinical outcomes in immune aplastic anemia. Blood. 2021 Dec 30;138(26):2799-2809. doi: 10.1182/blood.2021012895. PMID 34724566
- [Derived] Patel BA, Groarke EM, Lotter J, Shalhoub R, Gutierrez-Rodrigues F, Rios O, Quinones Raffo D, Wu CO, Young NS. Long-term outcomes in patients with severe aplastic anemia treated with immunosuppression and eltrombopag: a phase 2 study. Blood. 2022 Jan 6;139(1):34-43. doi: 10.1182/blood.2021012130. PMID 34525188
- [Derived] Zaimoku Y, Patel BA, Shalhoub R, Groarke EM, Feng X, Wu CO, Young NS. Predicting response of severe aplastic anemia to immunosuppression combined with eltrombopag. Haematologica. 2022 Jan 1;107(1):126-133. doi: 10.3324/haematol.2021.278413. PMID 33910334
- [Derived] Groarke EM, Patel BA, Gutierrez-Rodrigues F, Rios O, Lotter J, Baldoni D, St Pierre A, Shalhoub R, Wu CO, Townsley DM, Young NS. Eltrombopag added to immunosuppression for children with treatment-naive severe aplastic anaemia. Br J Haematol. 2021 Feb;192(3):605-614. doi: 10.1111/bjh.17232. Epub 2021 Jan 7. PMID 33410523
- [Derived] Giudice V, Wu Z, Kajigaya S, Fernandez Ibanez MDP, Rios O, Cheung F, Ito S, Young NS. Circulating S100A8 and S100A9 protein levels in plasma of patients with acquired aplastic anemia and myelodysplastic syndromes. Cytokine. 2019 Jan;113:462-465. doi: 10.1016/j.cyto.2018.06.025. Epub 2018 Jun 27. PMID 29958797
- [Derived] Giudice V, Banaszak LG, Gutierrez-Rodrigues F, Kajigaya S, Panjwani R, Ibanez MDPF, Rios O, Bleck CK, Stempinski ES, Raffo DQ, Townsley DM, Young NS. Circulating exosomal microRNAs in acquired aplastic anemia and myelodysplastic syndromes. Haematologica. 2018 Jul;103(7):1150-1159. doi: 10.3324/haematol.2017.182824. Epub 2018 Apr 19. PMID 29674506
- [Derived] Giudice V, Feng X, Lin Z, Hu W, Zhang F, Qiao W, Ibanez MDPF, Rios O, Young NS. Deep sequencing and flow cytometric characterization of expanded effector memory CD8+CD57+ T cells frequently reveals T-cell receptor Vbeta oligoclonality and CDR3 homology in acquired aplastic anemia. Haematologica. 2018 May;103(5):759-769. doi: 10.3324/haematol.2017.176701. Epub 2018 Feb 1. PMID 29419434
- [Derived] Hosokawa K, Muranski P, Feng X, Keyvanfar K, Townsley DM, Dumitriu B, Chen J, Kajigaya S, Taylor JG, Hourigan CS, Barrett AJ, Young NS. Identification of novel microRNA signatures linked to acquired aplastic anemia. Haematologica. 2015 Dec;100(12):1534-45. doi: 10.3324/haematol.2015.126128. Epub 2015 Sep 9. PMID 26354756
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-H-0150.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Recruitment has yet to be completed for the Extension Cohort, which was added to better assess the secondary endpoints
Groups:
- hATG, CsA, EPAG Day 14 to Month 6: Receive horse ATG days 1- 4, receive CsA day 1 to month 6, and receive eltrombopag day 14 to month 6
  hATG/CsA /eltrombopag -Cohort 1: hATG (standard of care) administered for 4 days, CsA (standard of care) administered starting day 1 for 6 months, eltrombopag (experimental) administered Day 14 to month 6
- hATG, CsA, EPAG Day 14 to Month 3: Receive horse ATG days 1- 4, receive CsA day 1 to month 6, and receive eltrombopag day 14 to month 3
  hATG/CsA /eltrombopag Cohort 2: hATG (standard of care) administered for 4 days, CsA (standard of care) administered starting day 1 for 6 months, eltrombopag (experimental) administered Day 14 to month 3
- hATG, CsA (Dose Reduced), EPAG Day 1 to Month 6: Receive horse ATG days 1- 4, receive CsA day 1 to month 6 at higher dose, then reduced dose for 18months, and receive eltrombopag day 1 to month 6
  hATG/CsA /eltrombopag Cohort 3: hATG (standard of care) administered for 4 days, CsA (standard of care) administered starting day 1 for 6 months at higher dose, then reduced dose for 18 months, eltrombopag (experimental) administered Day 1 to month 6
Period: Overall Study
Arm/Group | hATG, CsA, EPAG Day 14 to Month 6 | hATG, CsA, EPAG Day 14 to Month 3 | hATG, CsA (Dose Reduced), EPAG Day 1 to Month 6
Started | 30 | 31 | 31
Completed | 13 | 17 | 18
Not Completed | 17 | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hATG, CsA, EPAG Day 14 to Month 6 | hATG, CsA, EPAG Day 14 to Month 3 | hATG, CsA (Dose Reduced), EPAG Day 1 to Month 6 | Total
Number analyzed (Participants) | 30 | 31 | 31 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 8 | 19
  Between 18 and 65 years | 20 | 23 | 18 | 61
  >=65 years | 5 | 2 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 14 | 42
  Male | 16 | 17 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 9 | 17
  Not Hispanic or Latino | 24 | 29 | 22 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 4 | 16
  White | 16 | 19 | 23 | 58
  More than one race | 3 | 0 | 3 | 6
  Unknown or Not Reported | 3 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 31 | 92

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Hematologic Response
Description: Rate of complete hematologic response at six months for cohorts 1, 2 and 3.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | hATG, CsA, EPAG Day 14 to Month 6 | hATG, CsA, EPAG Day 14 to Month 3 | hATG, CsA (Dose Reduced), EPAG Day 1 to Month 6
Number analyzed (Participants) | 30 | 31 | 31
Participants
  No Response | 3 | 2 | 1
  Partial Response | 14 | 19 | 11
  Complete Response | 10 | 8 | 18
  Off study/Not Evaluable | 3 | 2 | 1

2. Secondary Outcome: Rate of Response at 3 and 12 Months Then Yearly; Rate of Relapse; Rate of Clonal Evolution to PNH, MDS and AML; Rate of Survival; Rate of Response for Relapse Subjects That Re-start Treatment and Effects of CsA Dose Starting at Month 6 to Month 24.
Description: Secondary endpoints will also be evaluated for the study to include: (a) hematological response at 3 and 12 months and yearly thereafter; (b) relapse (c) clonal evolution to PNH, clonal chromosomal population in bone marrow, myelodysplasia by morphology, or acute leukemia; (d) survival; (e) health-related quality of life; (f) hematological response of relapse subjects that re-start treatment; and (g) affects of a 2.0mg/kg/day CsA dose starting month 6 for 18 months until month 24 on the rate of relapse of subjects deemed responders at month 6.
Time Frame: 3 months to 5 years
Reporting Status: Not Posted, anticipated posting 2030-11

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | hATG, CsA, EPAG Day 14 to Month 6 | hATG, CsA, EPAG Day 14 to Month 3 | hATG, CsA (Dose Reduced), EPAG Day 1 to Month 6
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 17/30 | 15/31 | 14/31
Other Adverse Events (participants affected / at risk) | 30/30 | 31/31 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hATG, CsA, EPAG Day 14 to Month 6 (N=30) | hATG, CsA, EPAG Day 14 to Month 3 (N=31) | hATG, CsA (Dose Reduced), EPAG Day 1 to Month 6 (N=31)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (Red blood cells transfusion reaction) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 5 (8) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesophageal hernia, post elective laparascopic surgery (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (heel) (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (2) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Investigations) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycemia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ileal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune Hemolyitic Anemia Disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stenotrophomanas maltophilia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Sinusitis (Invasive Fungal Infection: Dematiaceous of nare/sinus) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas aeruginosa Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcus Epidermidis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Humerus and Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture, left (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Temperomandibular joint disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolisis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma, keratocantoma type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Volume overload (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 0 (0) | 2 (2) | 4 (4)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hATG, CsA, EPAG Day 14 to Month 6 (N=30) | hATG, CsA, EPAG Day 14 to Month 3 (N=31) | hATG, CsA (Dose Reduced), EPAG Day 1 to Month 6 (N=31)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 8 (17) | 11 (17)
Alanine aminotransferase increased (intermittent) (Investigations) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (4) | 7 (8)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 9 (10) | 9 (10) | 5 (8)
Blood bilirubin increased (intermittent) (Investigations) | 2 (3) | 4 (4) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis, intermittent (C. difficile) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid in the mastoid and inner ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Pressure behind ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye discoloration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Subconjunctival hemorrhage eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness transient (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
HSV mucositis: Mouth sore (aphthous ulcer) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gallstones (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3)
Hypokalemia (Investigations) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcus test positive (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Culture stool positive (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Smear cervix abnormal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleral disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic elastosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onychocryptosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Folliculitis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Debridement of nasal septum (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT01623167/Prot_SAP_000.pdf